CLINICAL TRIAL: NCT04173949
Title: Explorative Study for Treating Persistent Developmental Stuttering With Ramipril
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMC169-15
Record Dates: First submitted 2019-11-07; First posted 2019-11-22 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Persistent Developmental Stuttering
MeSH Terms: interventions — Ramipril

STUDY DESIGN:
Intervention Model Description: The study will begin as a pilot study in which 10 stuttering patients will be recruited for 12 weeks on open label Ramipril 2.5mg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ramipril 2.5 MG (Experimental): Ramipril 2.5 MG orall, daily.
  Interventions: Drug: Ramipril 2.5 MG

INTERVENTIONS:
Drug: Ramipril 2.5 MG — 3 month of treatment with daily Ramipril 2.5 MG

SUMMARY:
Persistent developmental stuttering (PDS) is diagnosed when developmental stuttering persists beyond adolescence. Most stutterers experience vast improvement in stuttering during childhood and it generally disappears within five years. A minority of stutterers continue stuttering over age 18, often accompanied by social and personal difficulties.

Following a report of a 75 year old woman, with severe Persistent developmental stuttering , who experienced significant improvement in her stuttering since treated by Ramipril for hypertension, we scrutinized the literature, and discovered that there is a physiological basis for this surprising reaction. Ace inhibitors, such as Ramipril, might in fact be successful for treating Persistent developmental stuttering .

In theory, it seems that ACE inhibitors, such as Ramipril could improve stuttering by reducing striatum dopamine levels.

1. Stuttering is associated with high striatum dopamine levels
2. Angiotensin receptors are present in the striatum
3. Angiotensin causes elevated striatum dopamine levels
4. ACE inhibitors penetrate the blood brain barrier and reduce brain angiotensin II levels.

Methods The study will begin as a pilot study in which 10 stuttering patients will be recruited for 12 weeks on open label Ramipril 1.25mg/d.

If there is improvement in at least 2 of the stuttering patients, we will continue to the main study.

Efficacy Evaluation:

1. The MINI Neuropsychiatric interview will be used to rule out major neuropsychiatric conditions
2. Stuttering evaluation

   1. Stuttering Severity instrument Version 4 (SSI-4) (Riley 2009)
   2. SLD :Percentage of stuttered syllables (Yairi 2015)
   3. The Subjective Screening of Stuttering (SSS)
   4. Speech Situation Checklist (Brutten 1975,1981)
3. Leibowitz Social Anxiety Scale (Leibowitz 1987)

The efficacy evaluation will be performed by speech therapists. All evaluations will be will be recorded on video

Safety evaluation:

1. Blood pressure: The average of three consecutive measures. Blood pressure will be measure in both arms on the first meeting, and thereafter on the arm with the highest measurements.
2. Orthostatic hypotension will be defined as a drop of 20mmHg systolic or 10mmHg diastolic, one and three minutes after standing from sitting position.
3. Creatinine clearance will be calculated by the MDRD method (Levy 2006) GFR, in mL/min per 1.73 m2 = 186.3 x SCr (exp[-1.154]) x Age (exp[-0.203]) x (0.742 if female) x (1.21 if black)

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Age 18 or above
* Developmental stuttering of 10 points severity at least (SSI-4)
* Agree not to have any speech or emotional therapy during the trial.

Exclusion Criteria:

* Systolic blood pressure < 110mmHg
* Estimated creatinine clearance < 50ml/min
* Baseline potassium > 5meq/ml
* Any sign of psychopathology by the MINI international neuropsychiatric interview
* Any psychotropic medications or substances in the past month
* History of angioedema or cough with any ACE inhibitor
* Aliskerin use in diabetes patients
* Current medication include ACE inhibitors or ARBS
* Pregnancy, or pregnancy plans during the study
* Less than 3% stuttered syllables
* Subjects with cluttering-stuttering when the cluttering is prominent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
changed in stuttered syllables | 4 month
  The difference in stuttering measures with and without treatment will be determined.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Haemek Medical Center, Afula
  - Asaf Harophe, Tzrifin

IPD SHARING:
Plan to Share IPD: No